CLINICAL TRIAL: NCT03393065
Title: Lung Ultrasound Guided Fluid Management Protocol for the Critically Ill Patient: a Randomized Study
Brief Title: Lung Ultrasound Guided Protocol for Fluid Management for the Critically Ill Patient: a Randomized Study
Acronym: LUNG US ICU
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Professor Adrian Covic (Other)
Responsible Party: Sponsor-Investigator, Professor Adrian Covic, Clinical Professor, Grigore T. Popa University of Medicine and Pharmacy
Organization: Grigore T. Popa University of Medicine and Pharmacy (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PN-III-P4-ID-PCE-2016-0908
Record Dates: First submitted 2017-12-06; First posted 2018-01-08 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Critical Illness
Keywords: lung ultrasounds; fluid managements; critical care patients
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Intervention Model Description: The patients will be randomized in two groups: in the intervention group pulmonary congestion, as assessed by the BLS will guide the fluid management, with a target of below 15 BLS. In the control group the fluid management will not be LUS guided. In both groups, further complementary fluid assessment methods will be performed blindly from the investigators: body composition assessment by bioimpedance and biochemical panel consisting in cardiac biomarkers (NTproBNP, cTnT) and inflamatory markers (IL-6).
Who Masked: Participant, Outcomes Assessor
Masking Description: Results of the lung ultrasounds will not be made publicly available
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group pulmonary congestion (Experimental): in the intervention group pulmonary congestion, as assessed by the BLS will guide the diuretic and fluid management, with a target of below 15 BLS. Furthermore, in the active arm, in the patients who will require a renal replacement therapy (RRT), BLS will be used to further guide the dialysis fluid prescription.
  Interventions: Other: Fluid management guided by BLS
- Control group (No Intervention): control group the fluid management will not be LUS guided

INTERVENTIONS:
Other: Fluid management guided by BLS — We propose a randomized study where in the interventional arm the fluid management (volume replacement, diuretics, use of vasopressors) will be guided using the BLS as a sign of pulmonary congestion.
  Arms: intervention group pulmonary congestion

SUMMARY:
In the Intensive Care Unit (ICU) this bedside method of assessing lung congestion could be useful in a better management of the critically ill patients with a wide range of respiratory failure causes (Acute Respiratory Distress Syndrome, COPD, acute pulmonary edema, pneumonia etc.). Fluid management is a key issue in the ICU where patients are either hemodynamic unstable and/or mechanically ventilated. A randomized study is proposed where in the interventional arm the fluid management (volume replacement, diuretics, use of vasopressors) will be guided using the BLS as a sign of pulmonary congestion.

DETAILED DESCRIPTION:
Inclusion criteria

- Age 18 or older admitted to the Intensive Care Unit

Exclusion criteria

* Due to LUS measurement limitation: patients with known persistent pleurisy, pulmonary fibrosis or pneumectomy;
* Unwillingness to participate in the study.

Active arm diuretic administration algorithm

* Intravenous diuretics will be used only to decrease the BLS to < 15;
* A stepped diuretic administration algorithm is provided below;
* Investigators may opt-out of the stepped diuretic administration algorithm if they feel it is in the best interests of the patient care;
* Intravenous diuretics can be decreased or temporarily discontinued if there is a decrease in blood pressure or an increase in creatinine that is felt to be due to a transient episode of intravascular volume depletion. After the patient has stabilized, if BLS ≥ 15, intravenous diuretics should be reinitiated until the patient's BLS is <15.

Active arm Initial BLS ≥ 15 Diuretic dose Previous Dose Suggested dose Furosemide (/day) Furosemide (/day) Hydrochlorothiazide (/day)

1. ≤ 80 mg 40 mg iv bolus + 5 mg/h 0
2. 81-160 mg 80 mg iv bolus + 10 mg/h 12.5 mg
3. 161-240 mg 80 mg iv bolus + 20 mg/h 25 mg
4. >240 mg 80 mg iv bolus + 30 mg/h 25 mg

At 24 hours Persistent BLS ≥ 15 Negative fluid balance > 1000 ml - reduce current diuretic regimen if desired Negative fluid balance < 1000 ml - maintain current diuretic regimen Positive fluid balance - advance to next step in table

Dialysis initiation AKI will be diagnosed based on changes in the serum creatinine, urine output, or both (according to the KDIGO recommendations). Creatinine measurements will be performed twice per day. Every patient will have a urinary catheter and urine output will be measured every hour.

Criteria for renal replacement therapy initiation:

Stage 3 AKI (urine output <0.3 mL/kg/h for ≥24 h and/or >3 fold increase in serum creatinine level compared with baseline or serum creatinine of ≥4 mg/dL with an acute increase of at least 0.5 mg/dL within 48 hours or

If any of the following absolute indications for RRT were present:

* Blood urea nitrogen level higher than 112 mg/dL;
* Serum potassium level higher than 6 mEq/L and/or with electrocardiography abnormalities;
* Urine production lower than 200 mL per 12 hours or anuria (according to the KDIGO recommendations);
* Organ edema in the presence of AKI resistant to diuretic treatment;
* A pH below 7.15 in the context of either pure metabolic acidosis (Paco2 below 35 mm Hg) or mixed acidosis (Paco2 of 50 mm Hg or more without the possibility of increasing alveolar ventilation)
* Acute pulmonary edema due to fluid overload responsible for severe hypoxemia requiring an oxygen flow rate greater than 5 liters per minute to maintain a Spo2 greater than 95% or requiring a Fio2 greater than 50% in patients receiving mechanical ventilation and despite diuretic therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older admitted to the Intensive Care Unit

Exclusion Criteria:

* known persistent pleurisy, pulmonary fibrosis or pneumectomy (due to lung ultrasonography limitations);
* unwillingness to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2017-12-01 (Actual); Primary Completion 2019-10-01 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
28 days survival | 28 days
  all-cause mortality

SECONDARY OUTCOMES:
Intensive care unit hospitalization | 28 days
  hospitalization in ICU
Duration of hospitalization | 28 days
  hospitalization
Days on mechanical ventilation | 28 days
  Need for mechanical ventilatory support

CONTACTS AND LOCATIONS:
Locations (1):
- Regional Institute of Oncology, Iasi, Iași, Romania

REFERENCES:
- [Background] Ciumanghel A, Siriopol I, Blaj M, Siriopol D, Gavrilovici C, Covic A. B-lines score on lung ultrasound as a direct measure of respiratory dysfunction in ICU patients with acute kidney injury. Int Urol Nephrol. 2018 Jan;50(1):113-119. doi: 10.1007/s11255-017-1730-8. Epub 2017 Oct 30. PMID 29086342
- [Derived] Rusu DM, Siriopol I, Grigoras I, Blaj M, Ciumanghel AI, Siriopol D, Nistor I, Onofriescu M, Sandu G, Cobzaru B, Scripcariu DV, Diaconu O, Covic AC. Lung Ultrasound Guided Fluid Management Protocol for the Critically Ill Patient: study protocol for a multi-centre randomized controlled trial. Trials. 2019 Apr 25;20(1):236. doi: 10.1186/s13063-019-3345-0. PMID 31023358